CLINICAL TRIAL: NCT04299737
Title: Improving Case Selection for Perioperative S. Aureus Transmission Surveillance to Reduce Surgical Site Infections
Status: Withdrawn | Type: Observational
Why Stopped: Due to the COVID-19 era, clinical research was interrupted, and this study was terminated.
Sponsor: Randy Loftus (Other)
Collaborators: RDB Bioinformatics (Industry)
Responsible Party: Sponsor-Investigator, Randy Loftus, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201911589
Record Dates: First submitted 2020-03-02; First posted 2020-03-09 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: S. Aureus Transmission

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First patient in the case pair: This patient will receive the treatment bundle. S. aureus transmission surveillance will be conducted.
  Interventions: Other: Treatment Bundle (as defined below)
- Second patient in the case pair: This patient will receive usual care. S. aureus transmission surveillance will be conducted.

INTERVENTIONS:
Other: Treatment Bundle (as defined below) — Patient decolonization within one hour of incision, improved environmental cleaning (frequency and quality, including but not limited to targeted use of no touch disinfection with UV-C treatment), provider hand hygiene leveraging proximity, improved catheter disinfection, and surveillance optimization.
  Groups: First patient in the case pair

SUMMARY:
The first patient in the dyad will receive the bundle, which includes patient decolonization methods, environmental cleaning in the OR, a hand hygiene system located on the IV pole for the anesthesia provider, and intravascular catheter and syringe tip disinfection practices. The second patient in the dyad will receive usual care. Both patients will be surveyed by obtaining swab samples at the beginning and end of the surgery using the OR PathTrac kits. The OR PathTrac software (RDB Bioinformatics, Omaha, NE 68154) uses algorithms to guide analysis of the S. aureus isolates and to identify transmission events. Transmission stories are processed by the software to generate transmission maps that identify improvement successes and failures. It also identifies actionable steps to improve the bundle. The perioperative infection control team then uses this information to continually optimize the bundle, and the software to measure the effect.

DETAILED DESCRIPTION:
Surgical site infections increase patient morbidity and healthcare costs. The Centers for Disease Control and Prevention emphasizes improved basic preventive measures to reduce bacterial transmission and infections for patients undergoing surgery.

Patients undergoing planned oncologic gynecological and plastic surgery will be entered as dyads into a worksheet each day that will rank and select the optimal cases. The research assistants consent both patients in the dyad to the study while they are in the Day of Surgery Admissions area. The first patient in the dyad will receive the bundle, which includes patient decolonization methods, environmental cleaning in the OR, a hand hygiene system located on the IV pole for the anesthesia provider, and intravascular catheter and syringe tip disinfection practices. The second patient in the dyad will receive usual care. Both patients will be surveyed by obtaining swab samples at the beginning and end of the surgery using the OR PathTrac kits. The OR PathTrac kits are obtained from and analyzed for S. aureus isolates by RDB Bioinformatics. The OR PathTrac software (RDB Bioinformatics, Omaha, NE 68154) uses algorithms to guide analysis of the S. aureus isolates and to identify transmission events. Transmission stories are processed by the software to generate transmission maps that identify improvement successes and failures. It also identifies actionable steps to improve the bundle. The perioperative infection control team then uses this information to continually optimize the bundle, and the software to measure the effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo oncologic gynecological and plastic surgery requiring general/regional anesthesia.
* informed, written consent.

Exclusion Criteria:

* Patients <18 years of age.
* Patients scheduled to undergo procedures outside of the surgical service lines listed above.
* Patients not requiring general or regional anesthesia.
* Patients who have a documented allergy or have an allergic reaction to to iodine, shellfish, or chlorhexidine.
* Patients who have not provided informed, written consent.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo oncologic gynecological and plastic surgery requiring general/regional anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Time course in S. aureus transmission decline with the intervention. | Up to 52 weeks
  S. aureus transmission events by time.

SECONDARY OUTCOMES:
Systematic selection of sequential cases in operating rooms for surveillance to reduce sample size and increase power. | Up to 52 weeks
  The outcome is the proportional reduction in the necessary sample size of pairs of cases achieved by systematic selection of sample cases as compared with random selection.

CONTACTS AND LOCATIONS:
Overall Officials: Randy W Loftus, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon written request and reviewed by the principal investigator for consideration.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon request and evaluation, if approved by the PI for release, at least one year from publication date.
Access Criteria: Submitted research protocol approved by the principal investigator, Dr. Loftus

REFERENCES:
- [Background] Loftus RW, Brown JR, Koff MD, Reddy S, Heard SO, Patel HM, Fernandez PG, Beach ML, Corwin HL, Jensen JT, Kispert D, Huysman B, Dodds TM, Ruoff KL, Yeager MP. Multiple reservoirs contribute to intraoperative bacterial transmission. Anesth Analg. 2012 Jun;114(6):1236-48. doi: 10.1213/ANE.0b013e31824970a2. Epub 2012 Mar 30. PMID 22467892
- [Background] Dexter F, Ledolter J, Epstein RH, Loftus RW. Importance of operating room case scheduling on analyses of observed reductions in surgical site infections from the purchase and installation of capital equipment in operating rooms. Am J Infect Control. 2020 May;48(5):566-572. doi: 10.1016/j.ajic.2019.08.017. Epub 2019 Oct 19. PMID 31640892
- [Background] Dexter F, Epstein RH, Gostine AL, Penning DH, Loftus RW. Benefit of systematic selection of pairs of cases matched by surgical specialty for surveillance of bacterial transmission in operating rooms. Am J Infect Control. 2020 Jun;48(6):682-687. doi: 10.1016/j.ajic.2019.09.025. Epub 2019 Nov 1. PMID 31679749
- [Background] Loftus RW, Koff MD, Brown JR, Patel HM, Jensen JT, Reddy S, Ruoff KL, Heard SO, Yeager MP, Dodds TM. The epidemiology of Staphylococcus aureus transmission in the anesthesia work area. Anesth Analg. 2015 Apr;120(4):807-18. doi: 10.1213/ANE.0b013e3182a8c16a. PMID 24937345
- [Background] German RR, Lee LM, Horan JM, Milstein RL, Pertowski CA, Waller MN; Guidelines Working Group Centers for Disease Control and Prevention (CDC). Updated guidelines for evaluating public health surveillance systems: recommendations from the Guidelines Working Group. MMWR Recomm Rep. 2001 Jul 27;50(RR-13):1-35; quiz CE1-7. PMID 18634202
- [Background] Rubin RH. Surgical wound infection: epidemiology, pathogenesis, diagnosis and management. BMC Infect Dis. 2006 Nov 27;6:171. doi: 10.1186/1471-2334-6-171. PMID 17129369
- [Background] Stulberg JJ, Delaney CP, Neuhauser DV, Aron DC, Fu P, Koroukian SM. Adherence to surgical care improvement project measures and the association with postoperative infections. JAMA. 2010 Jun 23;303(24):2479-85. doi: 10.1001/jama.2010.841. PMID 20571014
- [Background] Wang H, Hong S, Liu Y, Duan Y, Yin H. High inspired oxygen versus low inspired oxygen for reducing surgical site infection: a meta-analysis. Int Wound J. 2017 Feb;14(1):46-52. doi: 10.1111/iwj.12548. Epub 2015 Dec 23. PMID 26695819
- [Background] Koff MD, Loftus RW, Burchman CC, Schwartzman JD, Read ME, Henry ES, Beach ML. Reduction in intraoperative bacterial contamination of peripheral intravenous tubing through the use of a novel device. Anesthesiology. 2009 May;110(5):978-85. doi: 10.1097/ALN.0b013e3181a06ec3. PMID 19352154
- [Background] Loftus RW, Brindeiro BS, Kispert DP, Patel HM, Koff MD, Jensen JT, Dodds TM, Yeager MP, Ruoff KL, Gallagher JD, Beach ML, Brown JR. Reduction in intraoperative bacterial contamination of peripheral intravenous tubing through the use of a passive catheter care system. Anesth Analg. 2012 Dec;115(6):1315-23. doi: 10.1213/ANE.0b013e31826d2aa4. Epub 2012 Nov 9. PMID 23144441
- [Background] Phillips M, Rosenberg A, Shopsin B, Cuff G, Skeete F, Foti A, Kraemer K, Inglima K, Press R, Bosco J. Preventing surgical site infections: a randomized, open-label trial of nasal mupirocin ointment and nasal povidone-iodine solution. Infect Control Hosp Epidemiol. 2014 Jul;35(7):826-32. doi: 10.1086/676872. Epub 2014 May 21. PMID 24915210
- [Background] Loftus RW, Dexter F, Robinson ADM. High-risk Staphylococcus aureus transmission in the operating room: A call for widespread improvements in perioperative hand hygiene and patient decolonization practices. Am J Infect Control. 2018 Oct;46(10):1134-1141. doi: 10.1016/j.ajic.2018.04.211. Epub 2018 Jun 12. PMID 29907449
- [Background] Robinson ADM, Dexter F, Renkor V, Reddy S, Loftus RW. Operating room PathTrac analysis of current intraoperative Staphylococcus aureus transmission dynamics. Am J Infect Control. 2019 Oct;47(10):1240-1247. doi: 10.1016/j.ajic.2019.03.028. Epub 2019 Apr 27. PMID 31036398
- [Background] Durkin MJ, Dicks KV, Baker AW, Lewis SS, Moehring RW, Chen LF, Sexton DJ, Anderson DJ. Seasonal Variation of Common Surgical Site Infections: Does Season Matter? Infect Control Hosp Epidemiol. 2015 Sep;36(9):1011-6. doi: 10.1017/ice.2015.121. Epub 2015 May 26. PMID 26008876
- [Background] Munoz-Price LS, Bowdle A, Johnston BL, Bearman G, Camins BC, Dellinger EP, Geisz-Everson MA, Holzmann-Pazgal G, Murthy R, Pegues D, Prielipp RC, Rubin ZA, Schaffzin J, Yokoe D, Birnbach DJ. Infection prevention in the operating room anesthesia work area. Infect Control Hosp Epidemiol. 2019 Jan;40(1):1-17. doi: 10.1017/ice.2018.303. Epub 2018 Dec 11. No abstract available. PMID 30526699
- [Background] Schweizer ML, Chiang HY, Septimus E, Moody J, Braun B, Hafner J, Ward MA, Hickok J, Perencevich EN, Diekema DJ, Richards CL, Cavanaugh JE, Perlin JB, Herwaldt LA. Association of a bundled intervention with surgical site infections among patients undergoing cardiac, hip, or knee surgery. JAMA. 2015 Jun 2;313(21):2162-71. doi: 10.1001/jama.2015.5387. PMID 26034956
- [Background] Clark C, Taenzer A, Charette K, Whitty M. Decreasing contamination of the anesthesia environment. Am J Infect Control. 2014 Nov;42(11):1223-5. doi: 10.1016/j.ajic.2014.07.016. Epub 2014 Oct 30. PMID 25444268
- [Background] Wilson AP, Smyth D, Moore G, Singleton J, Jackson R, Gant V, Jeanes A, Shaw S, James E, Cooper B, Kafatos G, Cookson B, Singer M, Bellingan G. The impact of enhanced cleaning within the intensive care unit on contamination of the near-patient environment with hospital pathogens: a randomized crossover study in critical care units in two hospitals. Crit Care Med. 2011 Apr;39(4):651-8. doi: 10.1097/CCM.0b013e318206bc66. PMID 21242793
- [Background] Anderson DJ, Chen LF, Weber DJ, Moehring RW, Lewis SS, Triplett PF, Blocker M, Becherer P, Schwab JC, Knelson LP, Lokhnygina Y, Rutala WA, Kanamori H, Gergen MF, Sexton DJ; CDC Prevention Epicenters Program. Enhanced terminal room disinfection and acquisition and infection caused by multidrug-resistant organisms and Clostridium difficile (the Benefits of Enhanced Terminal Room Disinfection study): a cluster-randomised, multicentre, crossover study. Lancet. 2017 Feb 25;389(10071):805-814. doi: 10.1016/S0140-6736(16)31588-4. Epub 2017 Jan 17. PMID 28104287
- [Background] Loftus RW, Dexter F, Robinson ADM. Methicillin-resistant Staphylococcus aureus has greater risk of transmission in the operating room than methicillin-sensitive S aureus. Am J Infect Control. 2018 May;46(5):520-525. doi: 10.1016/j.ajic.2017.11.002. Epub 2018 Jan 4. PMID 29307750
- [Background] Loftus RW, Dexter F, Robinson ADM, Horswill AR. Desiccation tolerance is associated with Staphylococcus aureus hypertransmissibility, resistance and infection development in the operating room. J Hosp Infect. 2018 Nov;100(3):299-308. doi: 10.1016/j.jhin.2018.06.020. Epub 2018 Jun 30. PMID 29966756